CLINICAL TRIAL: NCT03252769
Title: Vaginal Self-sampling for High-risk HPV Detection in Women Who do Not Attend Cervical Screening
Brief Title: Vaginal Self-sampling for Non-attenders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Western Health and Social Care Trust (Other)
Responsible Party: Principal Investigator, Dr. Mary McMenamin, Dr., Western Health and Social Care Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: WT 15/15
Record Dates: First submitted 2017-08-15; First posted 2017-08-17 (Actual); Last update posted 2018-10-04 (Actual); Status verified 2018-10

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Self-sampling (Other): Invitation to self-sample
  Interventions: Other: Self-sampling

INTERVENTIONS:
Other: Self-sampling

SUMMARY:
Cervical cytology screening coverage in Northern Ireland (the proportion of eligible women, aged 25-64 years who have had a test result recorded in the previous five years) has increased steadily since 2005 to 78% in 2012/2013; almost reaching the 80% coverage target. The uptake of cervical screening among women in the 25-29 year age group in Northern Ireland however, has remained consistently lower (70-73%) than all other age groups except for the 60-64 year age group where the coverage rate is similar. The main barriers preventing women from attending for cervical screening are: embarrassment; inconvenience; time and discomfort associated with obtaining cervical samples. Studies have shown that offering women the opportunity to collect a vaginal self-sample to test for HPV (the main risk factor for cervical cancer) could increase screening coverage. Non-attenders in the Western and Belfast Health and Social Care Trust area, aged 25-29 years, will be identified by GPs. Letters with information relating to the study and collection devices will be sent to women giving them two options: 1. inviting them to book a normal screening appointment; 2. inviting them to collect a self-sample for HPV testing with either a swab or brush collection device. Participants for receipt of swab or brush will be randomised. Acceptance to participate in the study will be indicated by signed consent. Returned self-collected samples will be HPV tested. If a sample is negative, no further investigation is required and the woman will be encouraged to accept her next screening invitation. If a sample is positive the woman will be encouraged to book a screening appointment. The study will evaluate: impact on screening uptake, acceptance of self-sampling for both devices, practicality and cost-effectiveness of the intervention.

DETAILED DESCRIPTION:
Women aged 25-29 years who have not attended for cervical screening 9 months after being called initially will be considered non-attenders and therefore eligible participants. GPs will identify non-attenders and pass lists to cytology Audit Officers. A group of age-matched non-attenders will act as controls. Potential participants/controls will be ramdomly allocated to each group as cases arise. Study packs containing: invitation letters, participant information, consent forms and HPV self-sampling devices/instructions with return sample packaging will be sent to non-attenders, 3 months after their GP final reminder, by the Audit Officers inviting them to participate in the study by collecting a vaginal self-sample for HPV testing. The letter will contain two options for non-attenders: 1. inviting them to book a normal screening appointment (non-participation); 2. inviting them to participate in the study by collecting a self-sample for HPV testing with either a swab or brush collection device. Potential participants for receipt of swab or brush will be randomised. The participant information sheet will explain the purpose of the study, how the test is conducted, by the woman and at the laboratory, how the results will be conveyed to the woman and her GP and the implications of the HPV test result. The consent form will seek permission from the woman to process the sample, report the results to the woman, her GP and the screening office. In addition permission for the research team to check the patient LabCentre database for subsequent cervical screening results in the event of the woman testing HPV positive.

Women will return the self-sample to the Cytology laboratory, Altnaelvin in the pre-paid envelope provided. The sample will be HPV tested by the research team and the results sent to the woman, her GP and the screening office. Women who test HPV positive will be sent a results letter and advised to attend for cervical screening. The woman's GP will also be advised of the management recommendations. Women who test HPV positive will also be given a helpline number if they wish to discuss their result.

The research team will be responsible for recalling women who test HPV positive for cervical screening. A reminder letter will be sent to women who test HPV positive if they have not attended cervical screening 3 months post self-sampling intervention. Women who test HPV negative do not require further investigation so will be reassured and encouraged to accept their next screening invitation.

Women who have tested HPV positive but have negative cytology will be offered repeat HPV testing (GP collected sample) in 12 months and if this is still HPV positive the woman will be offered a further HPV test 12 months later. The research team will issue these invitations in conjunction with the woman's GP. Women with a persistent HPV infection will be referred to colposcopy by the research team.

The number of women returning the self-sampling devices and the number of HPV positive women attending for subsequent cervical screening will be monitored by the research team. The Audit Officers will provide anonymised cervical screening uptake data for control groups in order to ascertain the proportion of cervical screening samples that were obtained as a result of self-sampling/HPV positivity. Outcomes will be measured at 6 and 12 months post intervention result.

The study will last 18 months. The end of trial will be when the LabCentre database has been checked for cervical screening results obtained as a result of the intervention for all participants at the maximum time limit for return of self-samples plus 3 months to allow for return of HPV results to participants and recording of any cervical screening results on LabCentre.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 25-29y and 55-64y

Exclusion Criteria:

* Aged below 25y; between 30-54y or aged over 64y

Ages: 25 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1950 (Estimated)
Dates: Start 2016-05 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
The uptake rate of cervical screening in response to the intervention | 4 weeks - 6 months
  The uptake rate of cervical screening in response to the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Mary McMenamin, Principal Investigator — WHSCT
Locations (1):
- WHSCT, Londonderry, Northern Ireland, United Kingdom

IPD SHARING:
Plan to Share IPD: No